CLINICAL TRIAL: NCT04164628
Title: Investigation of Affecting Factors Quality of Life in Women
Brief Title: Evaluation of Quality of Life in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Arzu Demircioğlu, PT, Research Assisstant, MSc, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GO 19/1046
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Quality of Life; Women Health; Social Interaction
Keywords: quality of life; depression; anxiety; social function
MeSH Terms: conditions — Depression; Anxiety Disorders; Social Adjustment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group: quality of life assessment (Experimental): Women's quality of life will be evaluated.
  Interventions: Other: Quality of life assessment

INTERVENTIONS:
Other: Quality of life assessment — Quality of life will be assessed with Nottingham Health Profile

SUMMARY:
300 women will be evaluated in this study. Their quality of life, level of physical activity, Social Functioning, levels of depression and musculoskeletal status will be assessed.

DETAILED DESCRIPTION:
Many factors affects quality of life in women. In the literature, factors affecting the quality of life such as diseases, working conditions and psychological factors of women have been investigated in different diseases. However, there was no study investigating the factors affecting quality of life for a sample of adult female individuals. Therefore, the aim of our study is to investigate the effect of social, psychological and physical variables that we think may affect the quality of life in women.

ELIGIBILITY:
Inclusion Criteria:

* To be a volunteer

Exclusion Criteria:

* having severe musculoskeletal system disorders

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 227 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-28 (Actual)

PRIMARY OUTCOMES:
Quality of life | 5 minutes
  The Nottingham Health Profile is a general patient self-evaluation of subjective health status. The score of this questionnaire ranges between 0 and 600. The higher score indicates the worse quality of life.

SECONDARY OUTCOMES:
Social Functioning Scale | 10 minutes
  Questionnaire is specifically designed to assess the most relevant areas of social functioning. The higher score indicates the better social function.
Depression scale | 5 minutes
  The Beck Depression Inventory is a 21-item self-administered scale measuring various symptoms of depression. It comprises 21 groups of statements describing the somatic and cognitive-emotional symptoms of depression. Each item consists of four alternative responses.
  graded from 0 to 3 according to the severity of the symptom. The patients choose the response closest to their state during the past week. A sum score is counted, a higher score indicating more severe depression
physical activity level | 5 minutes
  Physical activity was assessed using the self-administered short (7-item) forms of the international physical activity questionnaire. The higher score indicates the more physically active lifestyle.
Musculoskeletal status | 5 minutes
  The Nordic musculoskeletal questionnaire includes 27 items exploring the presence of musculoskeletal symptoms during a 12-month period covering the nine different parts of the body. The higher score indicates the worse musculoskeletal status.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No